CLINICAL TRIAL: NCT01354457
Title: Evaluation of the Efficacy and Tolerance of Fractionated Radio-immunotherapy With 90Y-Epratuzumab (90Y-hLL2) for Relapsed or Refractory CD22+ B-Acute Lymphoblastic Leukaemia Patients
Brief Title: Safety and Efficacy of Radio-immunotherapy (RIT) for Patients With Relapse or Refractory Acute Lymphoblastic Leukaemia (ALL) B CD22+
Acronym: RIT 90YEpra
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 08/12-H
Record Dates: First submitted 2009-07-17; First posted 2011-05-16 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2011-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Patient with relapsing or refractory CD22+B-acute lymphoblastic leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epratuzumab and 90Y-Epratuzumab (Experimental): Escalating dose schedule with 5 cohort. For each cohort 3 patients will receive Radio-immunotherapy (RIT ) at Day 1 and Day 8 ± 2 First cohort : 92,5 MBq/m² of 90Y-DOTA-hLL2 associated with hLL2 Second cohort : 185 MBq/m² d'90Y-DOTA-hLL2 associated with hLL2 Third cohort : 277,5 MBq/m² d'90Y-DOTA-hLL2 associated with hLL2 Fourth cohort : 370 MBq/m² d'90Y-DOTA-hLL2 associated with hLL2 Fifth cohort : 462.5 MBq/m² d'90Y-DOTA-hLL2 associated with hLL2
  Interventions: Drug: Epratuzumab and 90Y-Epratuzumab

INTERVENTIONS:
Drug: Epratuzumab and 90Y-Epratuzumab — Sequential injections of each product with an escalating dose for radiolabeled Epratuzumab between patients

SUMMARY:
The purpose of this study is to determine whether fractionated RIT with Epratuzumab and radiolabeled Epratuzumab are effective in the treatment of relapsing or refractory ALL.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* B-ALL (OMS) with >=20% of blasts in bone marrow
* CD22+ expression >=70% of the blast population
* All previously treated ALL patients who have experienced relapse or treatment failure
* At least 15 days since previous treatment
* Performance status 0 - 2
* Creatinine clearance >= 50 ml/min (Cockroft formula).
* Serum bilirubin <= 30 mmol/l
* Written informed consent

Exclusion Criteria:

* T-ALL
* Meningeal involvement
* CD22 expression on tumor cells or < 70%
* HIV positive
* Active Hepatitis B or C
* Active infection within 7 days of starting treatment
* Left ventricular ejection fraction < 50%.
* Contra-indication to 90Y-DOTA-hLL2
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 5 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation at the same time in another study in which investigational drugs are used
* Absence of written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Determination of MTD by evaluation of hematological and non hematoligical toxicity
  The primary endpoint is to evaluate the incidence of dose limiting toxicities (DLT) in order to determine the maximal tolerated dose (MTD) in a dose escalating study design

SECONDARY OUTCOMES:
rate of haematological response
  To determine the hematologic response

CONTACTS AND LOCATIONS:
Overall Officials: Chevallier Patrice, MD, Principal Investigator — Nantes University Hospital; Kraeber-Bodere Françoise, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France

REFERENCES:
- [Derived] Chevallier P, Eugene T, Robillard N, Isnard F, Nicolini F, Escoffre-Barbe M, Huguet F, Hunault M, Marcais A, Gaschet J, Cherel M, Guillaume T, Delaunay J, Peterlin P, Eveillard M, Thomas X, Ifrah N, Lapusan S, Bodet-Milin C, Barbet J, Faivre-Chauvet A, Ferrer L, Bene MC, Le Houerou C, Goldenberg DM, Wegener WA, Kraeber-Bodere F. (90)Y-labelled anti-CD22 epratuzumab tetraxetan in adults with refractory or relapsed CD22-positive B-cell acute lymphoblastic leukaemia: a phase 1 dose-escalation study. Lancet Haematol. 2015 Mar;2(3):e108-17. doi: 10.1016/S2352-3026(15)00020-4. Epub 2015 Feb 25. PMID 26687796